CLINICAL TRIAL: NCT03738683
Title: Pharmacokinetics of Piperacillin and Tazobactam in Critically Ill Patients - Finding the Best Predictor for Piperacillin-tazobactam Clearance
Brief Title: Pharmacokinetics of Piperacillin and Tazobactam in Critically Ill Patients
Acronym: PICTAR
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Collaborators: UMC Utrecht (Other)
Responsible Party: Sponsor
Other Study IDs: UMCN-AKF 18.11
Record Dates: First submitted 2018-10-22; First posted 2018-11-13 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2019-09

CONDITIONS: Bacterial Infections
Keywords: Pharmacokinetics; Piperacillin-tazobactam; Renal function; Intensive Care Unit; Cystatin C
MeSH Terms: conditions — Bacterial Infections | interventions — Piperacillin, Tazobactam Drug Combination

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma samples for determination of total and free drug concentrations of piperacillin and tazobactam and for determination of cystatin C. Urine for measuring 24h creatinine clearance
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Piperacillin/tazobactam — Dose according to summary of product characteristics (SPC) or local protocols

SUMMARY:
Optimal understanding of piperacillin-tazobactam pharmacokinetics in critically ill patients is lacking resulting in large variation of achieved exposure and possible inadequate therapy. The investigators hypothesize that drug dosing based on CKD-EPIcr-cys provides a useful method to individualize and optimize therapy for piperacillin-tazobactam and eventually improve outcome.

In a multi-centre, observational, open-label study the investigators aim to define PK of free drug concentrations of both piperacillin and tazobactam in ICU patients and define a PK model for estimation of renal function that most accurately predicts piperacillin and tazobactam clearance.

DETAILED DESCRIPTION:
Infections in critically ill patients are a major healthcare problem and an important source of morbidity and mortality. Since critically ill patients often have altered pharmacokinetics (PK) compared to non-critically ill patients there is a substantial risk that present standard dosing regimens of antibiotics lead to suboptimal outcomes for patients on the ICU. To prevent the risk of inadequate dosing in ICU patients, it is important to fully understand the PK of antibiotics in this vulnerable group so that dosing regimens can be optimized.

Although PK of piperacillin has been well studied in healthy volunteers, non-critically ill patients and more recently the critically ill, there are still gaps of knowledge in the PK of piperacillin-tazobactam in ICU patients. Especially when focusing on the influence of renal function and on the PK of tazobactam.

Both piperacillin and tazobactam are excreted primarily by the kidneys via glomerular filtration and tubular secretion. Elimination half life of piperacillin-tazobactam increases with decreasing renal function. Substantial changes in renal function are common in ICU patients. Due to these changes PK targets are often not reached. This indicates the need to define the best predictor for piperacillin-tazobactam clearance in ICU patients in order to improve drug dosing. The use of combined filtration markers together, cystatin C and creatinine, can improve precision in estimating GFR (eGFR).

In a multi-centre, observational, open-label study the investigators aim to define PK of free drug concentrations of both piperacillin and tazobactam in ICU patients and define a PK model for estimation of renal function that most accurately predicts piperacillin and tazobactam clearance.

Patients will receive standard care, as stated in the product characteristics or according to local protocols. Minimally invasive blood sampling for pharmacokinetic analysis will be retrieved through a central venous catheter or an arterial line. Full pharmacokinetic curves will be taken for individual patients on the intermittent dosing regimen and limited sampling will be taken for individual patients on the continuous dosing regimen. A total of 40 patients will be included.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is admitted to an ICU.
2. Subject is at least 18 years old on the day of the first dosing.
3. Is managed with a central venous catheter or arterial line.
4. Patient is treated with piperacillin/tazobactam.

Exclusion Criteria:

1. Has previously participated in this trial.
2. Is on renal replacement therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All critically ill patients with a suspected or proven bacterial infection who are already treated with piperacillin-tazobactam as a part of routine clinical care are eligible for inclusion. A total of 40 patients will be included: 30 patients receiving intermittent infusion of piperacillin-tazobactam and 10 patients receiving continuous infusion.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Total drug clearance | 1 day
  Pharmacokinetic curves will be taken

SECONDARY OUTCOMES:
Volume of distribution | 1 day
  Pharmacokinetic curves will be taken
Area under the curve | 1 day
  Pharmacokinetic curves will be taken

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Radboud University Medical Center, Nijmegen, Gelderland
  - University Medical Centre Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wallenburg E, Ter Heine R, Schouten JA, Raaijmakers J, Ten Oever J, Kolwijck E, Burger DM, Pickkers P, Frenzel T, Bruggemann RJM. An Integral Pharmacokinetic Analysis of Piperacillin and Tazobactam in Plasma and Urine in Critically Ill Patients. Clin Pharmacokinet. 2022 Jun;61(6):907-918. doi: 10.1007/s40262-022-01113-6. Epub 2022 Apr 4. PMID 35377133